CLINICAL TRIAL: NCT00342004
Title: A Prospective Cohort Study of Occupational Exposures and Cancer Risk Among Women
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998006; OH98-C-N006
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer; Non-Hodgkin Lymphoma; Breast Cancer; Stomach Cancer; Brain Cancer
Keywords: Shanghai; Residential History; Exposure Assessment; Cohort Study; Molecular Epidemiology
MeSH Terms: conditions — Lung Neoplasms; Lymphoma, Non-Hodgkin; Breast Neoplasms; Stomach Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy female urban residents in Shanghai between ages of 40-70.

SUMMARY:
A prospective cohort study is proposed to evaluate occupational and environmental risk factors for cancer among women in Shanghai, China. Approximately 75,000 women aged 40-69 who reside in eight geographically defined communities in two urban districts of Shanghai will be recruited via a community-based cancer education program. All eligible subjects will be invited by local health workers from the neighborhood health station to the clinic for an interview and selected anthropometric measurements. The interview will elicit information on demographic background, diet, lifestyle factors, medical history, lifetime occupational history and residential history for the past 20 years. In addition, the women will be asked for information on their husbands' current and usual occupations, and demographic and a few other exposure factors. A spot urine sample and 10 ml of blood will be collected from all cohort members and stored at -70 degrees C for future assays of urine metabolites and DNA and hemoglobin adducts of selected occupational and environmental carcinogens, and polymorphic genes encoding enzymes that are involved in metabolism of relevant carcinogens. Cohort members and their husbands will be followed for cancer outcomes through biennial recontact and linkage with files of the population-based Shanghai Cancer Registry, of the Shanghai Vital Statistics, and of the Shanghai Resident Registry. Medical records and pathology slides will be reviewed for all cancer cases to verify their diagnosis. Post-diagnostic blood samples will be obtained from all cohort members diagnosed with cancer during the follow-up period and stored for future methodologic and etiologic studies. The proposed initial study period is 5 years, with an average follow-up of about 3.5 years. We anticipate, however, that follow-up will continue for 10 years or more.

DETAILED DESCRIPTION:
A prospective cohort study is proposed to evaluate occupational and environmental risk factors for cancer among women in Shanghai, China. Approximately 75,000 women aged 40-69 who reside in eight geographically defined communities in two urban districts of Shanghai will be recruited via a community-based cancer education program. All eligible subjects will be invited by local health workers from the neighborhood health station to the clinic for an interview and selected anthropometric measurements. The interview will elicit information on demographic background, diet, lifestyle factors, medical history, lifetime occupational history and residential history for the past 20 years. In addition, the women will be asked for information on their husbands' current and usual occupations, and demographic and a few other exposure factors. A spot urine sample and 10 ml of blood will be collected from all cohort members. Among participants who did not provide a blood sample, a buccal cell sample will be collected. All biological samples will be stored at -70 degrees C for future assays of genetic polymorphisms, urine metabolites and DNA and hemoglobin adducts of selected occupational and environmental carcinogenACs. Cohort members and their husbands will be followed for cancer outcomes through annual recontact and linkage with files of the population-based Shanghai Cancer Registry, of the Shanghai Vital Statistics, and of the Shanghai Resident Registry. Medical records and pathology slides will be reviewed for all cancer cases to verify their diagnosis. Post-diagnostic blood samples will be obtained from all cohort members diagnosed with cancer during the follow-up period and stored for future methodologic and etiologic studies. The proposed initial study period is 5 years, with an average follow-up of about 3.5 years. We anticipate, however, that follow-up will continue for 10 years or more.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women aged 40-69 who are permanent residents in eight geographically defined communities of urban Shanghai.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy female urban residents in Shanghai between ages of 40-70.
Sampling Method: Non-Probability Sample
Enrollment: 75366 (Actual)
Dates: Start 1997-05-01 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
All cancer incidence | up to 30 years
  Any cancer incidence, selected chronic diseases and all causemortality

SECONDARY OUTCOMES:
All deaths | up to 30 years
  All cause deaths

CONTACTS AND LOCATIONS:
Overall Officials: Qing Lan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Shanghai Cancer Institute, Shanghai, China

REFERENCES:
- [Background] Cantor KP, Stewart PA, Brinton LA, Dosemeci M. Occupational exposures and female breast cancer mortality in the United States. J Occup Environ Med. 1995 Mar;37(3):336-48. doi: 10.1097/00043764-199503000-00011. PMID 7796202
- [Background] Chow WH, Dosemeci M, Zheng W, Vetter R, McLaughlin JK, Gao YT, Blot WJ. Physical activity and occupational risk of colon cancer in Shanghai, China. Int J Epidemiol. 1993 Feb;22(1):23-9. doi: 10.1093/ije/22.1.23. PMID 8449643
- [Background] Chow WH, Ji BT, Dosemeci M, McLaughlin JK, Gao YT, Fraumeni JF Jr. Biliary tract cancers among textile and other workers in Shanghai, China. Am J Ind Med. 1996 Jul;30(1):36-40. doi: 10.1002/(SICI)1097-0274(199607)30:13.0.CO;2-Q. PMID 8837680